CLINICAL TRIAL: NCT02963571
Title: Posterior Percutaneous Pedicle Screw Fixation for Acute Thoracolumbar Vertebral Fractures With Simple Anterior Spinal Column Injury: a Retrospective, Self-controlled Trial
Brief Title: Posterior Percutaneous Pedicle Screw Fixation for Acute Thoracolumbar Vertebral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 153rd Hospital of Chinese People's Liberation Army (Other)
Responsible Party: Principal Investigator, Lei Liang, Attending Physician, 153rd Hospital of Chinese People's Liberation Army
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 153PLA_001
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Vertebral Fracture
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- screw fixation (Experimental): The patients underwent minimally invasive posterior percutaneous pedicle screw internal fixation.
  Interventions: Procedure: posterior percutaneous pedicle screw internal fixation

INTERVENTIONS:
Procedure: posterior percutaneous pedicle screw internal fixation — The patients underwent minimally invasive posterior percutaneous pedicle screw fixation in acute thoracolumbar vertebral fractures with simple anterior spinal column injury.

SUMMARY:
To validate the safety and effectiveness of minimally invasive posterior percutaneous pedicle screw fixation in acute thoracolumbar vertebral fractures with simple anterior spinal column injury.

DETAILED DESCRIPTION:
History and current related studies Thoracolumbar spinal fractures are frequently seen after trauma because of the biomechanical transitional junction of this structure. The primary treatment method used for traumatic thoracolumbar spinal fracture is posterior pedicle screw fixation, but this method has some disadvantages including severe trauma, extensive bleeding, long rehabilitation time, and long postoperative duration of intractable lumbar stiffness and low back pain. These complications occur mainly because of wide stripping and injury of the paraspinal muscles and peri-articular denervation. Percutaneous pedicle screw external fixation of spine fracture can reduce injury caused by screw insertion into the paraspinal muscles, particularly in the treatment of acute thoracolumbar vertebral compression fracture with simple anterior spinal column injury.

Adverse events We recorded possible adverse events, including wound pain, infection, back muscle pain, spinal cord/nerve injury, screw pull-out, or screw loosening. If severe adverse events occurred, details including the data of occurrence and measures taken to treat the adverse events were reported to the principle investigator and the institutional review board within 24 hours.

Possible biases and management measures Possible biases

* Diagnosis bias
* Admission rate bias (hospitalized patients were preferred to reduce loss to follow-up and to increase compliance)
* No response bias (subjects not responding to the questionnaire or not responding truthfully)
* Mixed bias (sex and age) Measures taken to control possible biases
* Formulation of strict inclusion and exclusion criteria
* Ensuring sample independence
* Discussion of the mixed factors that may potentially influence the curative effects, such as pathological factors, course of disease, and sex

Statistical analysis Statistical analysis was performed by a statistician using SPSS 19.0 software (IBM, Amrok, USA), and was conducted following the intention-to-treat principle. Normally distributed measurement data were expressed as the mean ± SD, and minimums and maximums. Non-normally distributed measurement data were expressed as lower quartile (q1), and median and upper quartile (q3). The Wilcoxon matched-pairs signed-ranks test was performed for comparison of the Cobb angle before surgery with the Cobb angle 3 years after surgery, and the McNemar's chi-squared test was used to compare the incidence of adverse reactions. The significance level was α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of acute thoracolumbar vertebral fracture with simple anterior spinal column injury as confirmed by radiography, CT and MRI
* AO classification type A
* Thoracolumbar injury severity score of 4-5 (Park et al., 2016)
* Traumatic fracture
* Age 25-47 years

Exclusion Criteria:

* Fracture complicated by spinal cord injury
* Fracture complicated by nerve injury
* Refusal to provide informed consent

Ages: 25 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The Cobb angle of the injured vertebral body | before, immediately after, and 3 months after surgery
  To investigate the change in the thoracolumbar spine curvature. A greater Cobb angle indicates more severe kyphosis.

SECONDARY OUTCOMES:
Anterior height of the injured vertebral body | before, immediately after, and 3 months after surgery
  To evaluate the morphological recovery of the thoracolumbar spine. A smaller anterior height of the injured vertebral body indicates less severe injury to the vertebral body.
X-ray | before, immediately after, and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lei Liang, Master, Principal Investigator — PLA 153 Central Hospital

IPD SHARING:
Plan to Share IPD: Undecided